CLINICAL TRIAL: NCT04935606
Title: mHealth to Enhance & Sustain Drug Use Reduction of the QUIT BI in Primary Care
Acronym: QUIT-Mobile
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Arkansas (Other); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Dallas Swendeman, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DA047386 (NIH); R01DA047386 (NIH)
Record Dates: First submitted 2020-10-07; First posted 2021-06-23 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Drug Use
Keywords: risky drug use; mobile phone; self-monitoring; automated feedback; SBIRT

STUDY DESIGN:
Intervention Model Description: 3-arm single blind RCT that compares: QUIT-Mobile, QUIT, and Usual Care, to assess the effectiveness among these interventions in reducing highest scoring risky drug use across time (at 3, 6 and 12 months follow-up).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Experimental): Usual Care participants will receive their standard medical care as usual (no provider advice or telephone coaching sessions) and all screening and study assessments. To reduce biases, Usual Care arm patients will be given a cancer screening booklet and will be shown a cancer screening Video Doctor. They will also receive 2 re-contact telephone sessions at weeks 2 and 6 corresponding to the timing of the coaching sessions for the QUIT and QUIT-Mobile arms. All participants will also receive re-contact calls monthly from 7-weeks to 12-months. The re-contact calls (5 min) provide attention control for the Usual Care arm, motivate continued trial participation by reminding them of the next research assessment, but do not provide an active intervention. At study end, the Usual Care arm will receive the QUIT video doctor and drug use reduction booklet brochure materials including overdose prevention materials and a list of clinic/community resources to help them reduce substance use.
  Interventions: Behavioral: Usual Care
- QUIT (Experimental): The QUIT brief intervention protocol will consist of 5 steps corresponding to the 5A's approach for assisting behavior change in the clinic setting (Ask, Advise, Assess, Assist, and Arrange) that will focus on patients' HSD (highest scoring drug on the baseline ASSIST) use in the past 30 days.
  Interventions: Behavioral: QUIT Intervention (doctor brief advice, video doctor, health coaching sessions at 2- and 6-weeks)
- QUIT-Mobile (Experimental): QUIT-Mobile will include a mobile platform with self-monitoring surveys and feedback message and robust data transfer protocols across three mobile technology platforms to meet diverse patient's preferences and needs regardless of literacy and phone type: a mobile-optimized web-app (using any smart phone's web-browser, not "native" apps), SMS (text-messaging), and IVR (automated voice calls for low literacy patients). Data collected during this study on patient platform preferences and exploratory analyses on intervention efficacy across platform types will inform the development of future effectiveness trials that can evaluate effectiveness of different mobile platforms.
  Interventions: Behavioral: QUIT-Mobile (QUIT Intervention plus weekly mobile-web app or text message weekly self-monitoring, automated feedback over 12 months)

INTERVENTIONS:
Behavioral: Usual Care — Usual Care participants will receive their standard medical care as usual and all study assessments. Providers will not receive information about their drug use. To reduce Hawthorne effect biases and to mask the study's purpose, RAs will provide the Usual Care arm patients with a cancer screening booklet and have them view a cancer screening Video Doctor. Participants will receive re-contact calls (5 min) to provide attentional control for the Usual Care arm, motivate continued trial participation by reminding next research assessment and study incentives, update contact information, and address participation barriers, but do not provide intervention. At study end, Usual Care will receive the QUIT video doctor and drug use reduction booklet materials including overdose prevention materials and a list of clinic/community resources to help them reduce substance use.
  Arms: Usual Care
Behavioral: QUIT Intervention (doctor brief advice, video doctor, health coaching sessions at 2- and 6-weeks) — QUIT's core components include:
  1. patient screening with the WHO Alcohol Smoking and Substance Involvement Screening Test (ASSIST, score 4-26);
  2. face-to-face brief clinician advice on reducing drug use (2-3 minutes);
  3. video doctor reinforcing the clinician message;
  4. drug use reduction brochure;
  5. 2- and 6-week telephone health coaching sessions to enhance self-efficacy in reducing drug use, via motivational interviewing and cognitive behavior therapy (CBT) techniques (20-30 minutes).
  Arms: QUIT
Behavioral: QUIT-Mobile (QUIT Intervention plus weekly mobile-web app or text message weekly self-monitoring, automated feedback over 12 months) — The QUIT-Mobile intervention includes QUIT's core components and adds:
  1. SMS/IVR/mobile-app self-monitoring survey prompts twice-weekly during the QUIT coaching through 6 weeks, and then weekly self-monitoring and automated feedback via SMS/IVR/app through 12-months.
  2. Web-based dashboards will be used by coaches for monitoring of patients' self-monitoring data to enhance 2- and 6-week coaching sessions and for monitoring during the post-coaching self-management and monitoring period from 7-weeks to 12-months and intervening accordingly. The mobile platform will provide the same intervention functions (self-monitoring surveys and feedback messages) and robust data transfer protocols across three mobile technology platforms.
  Arms: QUIT-Mobile

SUMMARY:
The QUIT-Mobile study proposes to use mobile phone self-monitoring and feedback to enhance and sustain over 12-months the impacts of the Quit Using Drugs Intervention Trial (QUIT), an effective screening and brief intervention (SBI) previously successful in reducing risky drug use (i.e., moderate use) in low-income, diverse patients over a 3-month follow up. The investigators will conduct the QUIT-Mobile study for patients who receive care in clinics of federally qualified health centers (FQHC) in Southern California over 12-months follow up. The study is an Effectiveness-Implementation Hybrid Type 1 design consisting of a single-blind, 3-arm, RCT with adult, mostly Latino FQHC primary care patients with risky drug use (ASSIST score 4-26), randomized to 3 conditions (n=200/arm, n=600 total): 1) QUIT-Mobile; 2) standard QUIT; 3) Usual Care. Qualitative data on implementation facilitators and barriers will inform future scale-up and sustainability, in addition to cost data analyses. The aims are to examine effectiveness in reducing risky drug use and cost-effectiveness comparing the three arms over 3-, 6- and 12-months. Drug use measures include self-reports for past 30-days and urine drug screen validation for underreporting (acknowledging that people with moderate risk drug use have sporadic drug use patterns requiring longer self-report recalls for drug use that urine screens may not detect). The 3-arm study enables testing of the independent and synergistic effects of QUIT-Mobile compared to QUIT and both to Usual Care. The 12-month timeline reflects annual primary care visits when screening and brief intervention would be repeated routinely. The QUIT intervention contains 3 primary components: 1) patient screening with the WHO ASSIST, 2) brief clinician advice (<3 minutes) including opioid overdose prevention education, and 3) 2- and 6-week telephone drug-use health coaching sessions utilizing motivational interviewing and cognitive behavioral techniques, delivered by paraprofessional health coaches. QUIT-Mobile tests the addition of mobile phone self-monitoring, automated feedback, and coach monitoring dashboard to enhance and sustain QUIT's drug use reductions using mobile-web app, text-messaging (SMS), or interactive voice response (IVR).

DETAILED DESCRIPTION:
The US Mental Health Parity Act encourages primary care (PC) providers to integrate behavioral health, including drug use reduction, into routine PC. QUIT (the Quit Using Drugs Intervention Trial), a multi-component screening and brief intervention (SBI) for diverse drug using adults in PC, reduces risky drug use and improves quality of life (QoL) over 3 months; the findings have been replicated in a subsequent study. Three key evidence gaps are: a) the effectiveness of SBI for people with moderate risk drug use over 6- and 12-months; b) low-cost methods to enhance, sustain, and monitor drug use reductions; and c) implementation barriers, facilitators, and costs of SBI for people with moderate risk drug use in PC. This study is an Effectiveness-Implementation Hybrid Type 1 design consisting of a 3-arm RCT and qualitative research.

QUIT is a four-pronged program: 1) patient screener at reception via tablet-device; 2) brief clinician advice (<5-minute); 3) video doctor reinforcing clinician advice; and 4) two telephone health coaching calls at 2- & 6-weeks. Mobile phone "apps," text-messaging (SMS), and interactive voice response (IVR) tools offer opportunities to enhance, sustain, and monitor effects of SBIs by facilitating patient activation and self-management between coaching sessions during daily routines, and sustaining changes after coaching ends.

QUIT-Mobile augments QUIT with 3 key functions: 1) patient self-monitoring of drug use and related factors (i.e., cravings, pain, physical and mental health symptoms/QoL) twice weekly by app, SMS, or IVR (per patient preference) and weekly from 6 wks to 12mo; 2) weekly automated feedback on goal progress for reducing drug use; and 3) dashboards for coach monitoring of patients' self-monitoring data. These functions aim to: enhance coaching sessions by facilitating goal tracking, problem solving, and patient-coach engagement; and after coaching to sustain patient activation; and monitor patients to prompt coach follow-up if drug use increases.

Self-monitoring is a core element of self-regulation and self-management applied in a range of chronic conditions. SMS, IVR, and apps enable self-monitoring and automated feedback to be cheaply implemented and scaled. The theoretical bases underlying QUIT's cognitive behavioral and motivational interviewing strategies emphasize that self-monitoring and feedback are integral to self-regulation and self-management through self-observation, reflection, self-correction, and reinforcement via self-reward, critique, and feedback.

Effectiveness of QUIT-Mobile and QUIT over 12-months will be examined in a single-blind, 3- arm, RCT with low-income, adult, mainly ethnic minority FQHC PC patients with risky drug use (RDU - based on ASSIST score 4-26; ASAM level 0.5), randomized to 3 conditions (n=200/arm, 600 total): 1) QUIT-Mobile, 2) standard QUIT, and 3) Usual Care (UC). Primary outcomes are drug use reductions measured by self-reports of past 30 days drug use (due to sporadic use patterns of people with moderate/risky drug use) with urine screen validation measured at baseline, 3-, 6-, and 12-months. Subgroups will be compared on outcomes by demographics, drug type, intervention engagement, comorbidities, pain, and clinic-level factors. Secondary outcomes are health services utilization and quality of life. Formative Qualitative Research will be conducted with patients, coaches, FQHC staff (providers, administrators, executives), payers / insurers and policy stakeholders to identify barriers/facilitators to adoption, implementation and sustainability. The Consolidated Framework for Implementation Research (CFIR) will guide this work. Costs will also be monitored, and cost analyses will be conducted.

Study Outcomes:

Primary: Reductions in use of the highest scoring drug on the ASSIST at baseline (that was used in the past 30 days) across time at 3-, 6- and 12- months follow-up, as measured by number of days of drug use in the past 30 days.

Secondary: 1) Improvement of quality of life as measured by the SF-12 physical and mental health scores; 2) costs analyses of the interventions for reducing drug use, including use of health services utilization data from EHR reviews; 3) barriers and facilitators to intervention implementation from qualitative reports with providers and clinic stakeholder, patients, and payer and policy maker stakeholders; 4) drug use reductions measured by timeline follow back (TLFB) of past 30 days use.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and older receiving care at study clinics.
* Have a phone number at which they can be contacted over time during the study (to conduct follow-up health education phone calls).
* Have a primary care visit with a regular clinic provider on the date of recruitment and enrollment.
* English or Spanish-speaking.
* ASSIST score between 4 and 26 indicating risky (moderate) drug use, and used the substance in the past 30 days.
* Able (not cognitively impaired) and willing to cooperate with data collection and research procedures, including and 2-week, 6-week, and 3, 6, 12-month follow-up assessments.
* Planning to be in the Los Angeles area for the next 12 months so they can complete the study period.

Exclusion Criteria:

* Pregnancy: Women who report being pregnant at the time of randomization will be excluded from participation. This latter exclusion criterion is based on the following reasons: (a) The interaction of drug use (in any amount) and fetal-maternal health is physiologically complex and beyond the scope of this proposed intervention. (b) Drug users who are pregnant are considered high-risk pregnancies.
* Repeaters: All patients will be asked a set of repeater questions. This includes a question on whether they have ever been involved in our UCLA study at the clinic before. We will create a unique identifier based on a set of questions that we have used in our prior studies that combines aspects about the potential subject (mother's first name, father's first name, month and day of birth) that will screen them out if they screen again in the future.
* ASSIST Score above 26 indicating high use and potential serious SUD needing referral to specialty treatment: The RA will receive a message that the subject scored 27+ on alcohol or any drugs on the WHO ASSIST (i.e. indication of possible severe substance use disorder). The RA will inform the patient that they are at risk for certain health behaviors and ask the patient if they want to disclose this information to their doctor. If they agree to disclose information to their doctor then we will fill out a letter informing the doctor of patient's potential more serious substance use disorder. We will also provide the patient with a list of local substance use disorder treatment referrals.
* ASSIST Score below 4 (low use): These patients are not eligible for enrollment in the trial.
* Subject Enrolled in a Substance Use Treatment Program: Subjects enrolled in a treatment program are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Drug Use | Baseline
  30-day self-reports of drug use (due to sporadic use patterns of moderate/risky drug users) with urine screen to validate underreporting given detection windows of 1-3 days for most drugs (except cannabis) measured at baseline.
Drug Use | 3-month follow-up
  30-day self-reports of drug use (due to sporadic use patterns of moderate/risky drug users) with urine screen to validate underreporting given detection windows of 1-3 days for most drugs (except cannabis) measured at 3-month follow-up.
Drug Use | 6-month follow-up
  30-day self-reports of drug use (due to sporadic use patterns of moderate/risky drug users) with urine screen to validate underreporting given detection windows of 1-3 days for most drugs (except cannabis) measured at 6-month follow-up.
Drug Use | 12-month follow-up
  30-day self-reports of drug use (due to sporadic use patterns of moderate/risky drug users) with urine screen to validate underreporting given detection windows of 1-3 days for most drugs (except cannabis) measured at 12-month follow-up.

SECONDARY OUTCOMES:
Health-related Quality of Life Improvement Self-Reports (SF-12) | Baseline
  Mental health status/QoL (SF-12):
  i. Physical Functioning: [1=Yes, Limited A Lot; 3= No, Not Limited At All] ii. Role- Physical: [1=Yes; 2=No] iii. Bodily Pain: [1=Not At All; 5=Extremely] iv. General Health: [1=Excellent; 5=Poor] v. Vitality: [1=All of the Time; 6=None of the Time] vi. Social Functioning: [1=All of the Time; 6=None of the Time] vii. Role- Emotional: [1=Yes; 2=No] viii. Mental Health [1=All of the Time; 6=None of the Time]
Health-related Quality of Life Improvement Self-Reports (SF-12) | 3-month follow-up
  Mental health status/QoL (SF-12):
  i. Physical Functioning: [1=Yes, Limited A Lot; 3= No, Not Limited At All] ii. Role- Physical: [1=Yes; 2=No] iii. Bodily Pain: [1=Not At All; 5=Extremely] iv. General Health: [1=Excellent; 5=Poor] v. Vitality: [1=All of the Time; 6=None of the Time] vi. Social Functioning: [1=All of the Time; 6=None of the Time] vii. Role- Emotional: [1=Yes; 2=No] viii. Mental Health [1=All of the Time; 6=None of the Time]
Health-related Quality of Life Improvement Self-Reports (SF-12) | 6-month follow-up
  Mental health status/QoL (SF-12):
  i. Physical Functioning: [1=Yes, Limited A Lot; 3= No, Not Limited At All] ii. Role- Physical: [1=Yes; 2=No] iii. Bodily Pain: [1=Not At All; 5=Extremely] iv. General Health: [1=Excellent; 5=Poor] v. Vitality: [1=All of the Time; 6=None of the Time] vi. Social Functioning: [1=All of the Time; 6=None of the Time] vii. Role- Emotional: [1=Yes; 2=No] viii. Mental Health [1=All of the Time; 6=None of the Time]
Health-related Quality of Life Improvement Self-Reports (SF-12) | 12-month follow-up
  Mental health status/QoL (SF-12):
  i. Physical Functioning: [1=Yes, Limited A Lot; 3= No, Not Limited At All] ii. Role- Physical: [1=Yes; 2=No] iii. Bodily Pain: [1=Not At All; 5=Extremely] iv. General Health: [1=Excellent; 5=Poor] v. Vitality: [1=All of the Time; 6=None of the Time] vi. Social Functioning: [1=All of the Time; 6=None of the Time] vii. Role- Emotional: [1=Yes; 2=No] viii. Mental Health [1=All of the Time; 6=None of the Time]
Health-related Quality of Life Improvement Self-Reports (MHI) | Baseline
  Two additional mental health questions will be collected at baseline, 3-, 6-, and 12-months follow-ups using the Mental Health Inventory (MHI) survey :
  i. "How much of the time during the past 4 weeks:" Have you been a very nervous person? [1=All of the Time; 6=None of the Time] Have you felt so down in the dumps that nothing could cheer you up? [1=All of the Time; 6=None of the Time]
Health-related Quality of Life Improvement Self-Reports (MHI) | 3-month follow-up
  Two additional mental health questions will be collected at baseline, 3-, 6-, and 12-months follow-ups using the Mental Health Inventory (MHI) survey :
  i. "How much of the time during the past 4 weeks:" Have you been a very nervous person? [1=All of the Time; 6=None of the Time] Have you felt so down in the dumps that nothing could cheer you up? [1=All of the Time; 6=None of the Time]
Health-related Quality of Life Improvement Self-Reports (MHI) | 6-month follow-up
  Two additional mental health questions will be collected at baseline, 3-, 6-, and 12-months follow-ups using the Mental Health Inventory (MHI) survey :
  i. "How much of the time during the past 4 weeks:" Have you been a very nervous person? [1=All of the Time; 6=None of the Time] Have you felt so down in the dumps that nothing could cheer you up? [1=All of the Time; 6=None of the Time]
Health-related Quality of Life Improvement Self-Reports (MHI) | 12-month follow-up
  Two additional mental health questions will be collected at baseline, 3-, 6-, and 12-months follow-ups using the Mental Health Inventory (MHI) survey :
  i. "How much of the time during the past 4 weeks:" Have you been a very nervous person? [1=All of the Time; 6=None of the Time] Have you felt so down in the dumps that nothing could cheer you up? [1=All of the Time; 6=None of the Time]
Health-related Quality of Life Improvement Self-Reports (WHOQoLBREF) | Baseline
  Insomnia (WHOQoLBREF) as assessed by, "Do you have any difficulties with sleeping?" [1=Not at all; 5=An extreme amount]
Health-related Quality of Life Improvement Self-Reports (WHOQoLBREF) | 3-month follow-up
  Insomnia (WHOQoLBREF) as assessed by, "Do you have any difficulties with sleeping?" [1=Not at all; 5=An extreme amount]
Health-related Quality of Life Improvement Self-Reports (WHOQoLBREF) | 6-month follow-up
  Insomnia (WHOQoLBREF) as assessed by, "Do you have any difficulties with sleeping?" [1=Not at all; 5=An extreme amount]
Health-related Quality of Life Improvement Self-Reports (WHOQoLBREF) | 12-month follow-up
  Insomnia (WHOQoLBREF) as assessed by, "Do you have any difficulties with sleeping?" [1=Not at all; 5=An extreme amount]
Health Service Utilizations | Baseline
  Health services utilization self-reports using 6- and 12-month recall periods of: # ED visits, # hospitalizations, # hospital days, # and type of outpatient visits. Self-reports are valid for 12-month recall. Electronic Health Records will be reviewed for additional data.
Health Service Utilizations | 3-month follow-up
  Health services utilization self-reports using 6- and 12-month recall periods of: # ED visits, # hospitalizations, # hospital days, # and type of outpatient visits. Self-reports are valid for 12-month recall. Electronic Health Records will be reviewed for additional data.
Health Service Utilizations | 6-month follow-up
  Health services utilization self-reports using 6- and 12-month recall periods of: # ED visits, # hospitalizations, # hospital days, # and type of outpatient visits. Self-reports are valid for 12-month recall. Electronic Health Records will be reviewed for additional data.
Health Service Utilizations | 12-month follow-up
  Health services utilization self-reports using 6- and 12-month recall periods of: # ED visits, # hospitalizations, # hospital days, # and type of outpatient visits. Self-reports are valid for 12-month recall. Electronic Health Records will be reviewed for additional data.
30-day Timeline Follow Back (TLFB) of Drug Use | Baseline
  TLFB will be assessed by including a calendar in the study web application where participants will click each day they used their highest scoring drug. Reported use on each day is then summed to achieve a summary score for the total number of days that drugs were used.
30-day Timeline Follow Back (TLFB) of Drug Use | 3-month follow-up
  TLFB will be assessed by including a calendar in the study web application where participants will click each day they used their highest scoring drug. Reported use on each day is then summed to achieve a summary score for the total number of days that drugs were used.
30-day Timeline Follow Back (TLFB) of Drug Use | 6-month follow-up
  TLFB will be assessed by including a calendar in the study web application where participants will click each day they used their highest scoring drug. Reported use on each day is then summed to achieve a summary score for the total number of days that drugs were used.
30-day Timeline Follow Back (TLFB) of Drug Use | 12-month follow-up
  TLFB will be assessed by including a calendar in the study web application where participants will click each day they used their highest scoring drug. Reported use on each day is then summed to achieve a summary score for the total number of days that drugs were used.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Gelberg, MD, MSPH, Principal Investigator — University of California, Los Angeles; Dallas Swendeman, PhD, MPH, Principal Investigator — University of California, Los Angeles
Locations (5):
- United States (5):
  - The Children's Clinic (TCC) Family Health, Long Beach, California
  - South Central Family Health Clinic, Los Angeles, California
  - Wesley Health Centers, Los Angeles, California
  - Saban Community Clinic, Los Angeles, California
  - UMMA Community Clinic, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a data sharing platform (to be determined) and upon request to PIs
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Background] Swendeman D, Sumstine S, Aguilar E, Gorbach PM, Comulada WS, Gelberg L. Feasibility and Acceptability of Mobile Phone Self-monitoring and Automated Feedback to Enhance Telephone Coaching for People With Risky Substance Use: The QUIT-Mobile Pilot Study. J Addict Med. 2021 Apr 1;15(2):120-129. doi: 10.1097/ADM.0000000000000707. PMID 32732684
- [Background] Gelberg L, Andersen RM, Afifi AA, Leake BD, Arangua L, Vahidi M, Singleton K, Yacenda-Murphy J, Shoptaw S, Fleming MF, Baumeister SE. Project QUIT (Quit Using Drugs Intervention Trial): a randomized controlled trial of a primary care-based multi-component brief intervention to reduce risky drug use. Addiction. 2015 Nov;110(11):1777-90. doi: 10.1111/add.12993. PMID 26471159
- [Background] Singleton KW, Lan M, Arnold C, Vahidi M, Arangua L, Gelberg L, Bui AA. Wireless data collection of self-administered surveys using tablet computers. AMIA Annu Symp Proc. 2011;2011:1261-9. Epub 2011 Oct 22. PMID 22195187
- [Background] Baumeister SE, Gelberg L, Leake BD, Yacenda-Murphy J, Vahidi M, Andersen RM. Effect of a primary care based brief intervention trial among risky drug users on health-related quality of life. Drug Alcohol Depend. 2014 Sep 1;142:254-61. doi: 10.1016/j.drugalcdep.2014.06.034. Epub 2014 Jul 4. PMID 25042213
- [Background] Bone C, Gelberg L, Vahidi M, Leake B, Yacenda-Murphy J, Andersen RM. Under-reporting of Risky Drug Use Among Primary Care Patients in Federally Qualified Health Centers. J Addict Med. 2016 Nov/Dec;10(6):387-394. doi: 10.1097/ADM.0000000000000246. PMID 27753718
- [Background] Reddy AT, Andersen RM, Gelberg L. Clinicians' Beliefs and Practices Regarding Drug Use Care of Their Community Health Center Patients. J Addict Med. 2015 Nov-Dec;9(6):447-53. doi: 10.1097/ADM.0000000000000158. PMID 26441402
- [Background] Padwa H, Ni YM, Barth-Rogers Y, Arangua L, Andersen R, Gelberg L. Barriers to drug use behavior change among primary care patients in urban United States community health centers. Subst Use Misuse. 2014 May;49(6):743-51. doi: 10.3109/10826084.2013.866962. Epub 2013 Dec 20. PMID 24354547
- [Background] Bone CW, Goodfellow AM, Vahidi M, Gelberg L. Prevalence of Sexual Violence and its Association with Depression among Male and Female Patients with Risky Drug Use in Urban Federally Qualified Health Centers. J Urban Health. 2018 Feb;95(1):111-115. doi: 10.1007/s11524-017-0213-7. PMID 29340911
- [Background] Gelberg L, Andersen RM, Rico MW, Vahidi M, Natera Rey G, Shoptaw S, Leake BD, Serota M, Singleton K, Baumeister SE. A pilot replication of QUIT, a randomized controlled trial of a brief intervention for reducing risky drug use, among Latino primary care patients. Drug Alcohol Depend. 2017 Oct 1;179:433-440. doi: 10.1016/j.drugalcdep.2017.04.022. Epub 2017 Jun 13. PMID 28844733
- [Background] Gelberg L, Natera Rey G, Andersen RM, Arroyo M, Bojorquez-Chapela I, Rico MW, Vahidi M, Yacenda-Murphy J, Arangua L, Serota M. Prevalence of Substance Use Among Patients of Community Health Centers in East Los Angeles and Tijuana. Subst Use Misuse. 2017 Feb 23;52(3):359-372. doi: 10.1080/10826084.2016.1227848. Epub 2016 Dec 21. PMID 28001094